CLINICAL TRIAL: NCT03818516
Title: Impact of Inflammation on Reward Circuits, Motivational Deficits and Negative Symptoms in Schizophrenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, David Goldsmith, Assistant Professor, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: IRB00094972; 1K23MH114037-01A1 (NIH)
Record Dates: First submitted 2019-01-19; First posted 2019-01-28 (Actual); Results first posted 2024-05-02 (Actual); Last update posted 2024-05-02 (Actual); Status verified 2024-04

CONDITIONS: Schizophrenia
Keywords: Inflammation; Magnetic Resonance Imaging (MRI); Negative Symptoms
MeSH Terms: conditions — Schizophrenia; Inflammation | interventions — Glucose Tolerance Test

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Oral Glucose Tolerance Test (OGTT) (Experimental): Medically stable participants with schizophrenia and a range of insulin resistance will have an oral glucose tolerance test.
  Interventions: Other: Oral Glucose Tolerance Test (OGTT)

INTERVENTIONS:
Other: Oral Glucose Tolerance Test (OGTT) — Participants will undergo a fasting blood draw for inflammatory and metabolic markers before a 75gm oral glucose tolerance test (OGTT) and at 1, 2 and 3 hours post-OGTT. Behavioral assessments will also be administered pre- and post-OGTT administration.

SUMMARY:
This study will recruit persons with schizophrenia or schizoaffective disorder and will use an oral glucose tolerance test to test the hypothesis that insulin resistance drives inflammation.

DETAILED DESCRIPTION:
Schizophrenia is a severe mental illness that affects 1% of the population, but accounts for over $60 billion in costs to the national healthcare system. Negative symptoms of schizophrenia, including motivational deficits, are some of the most debilitating aspects of the disorder, being both difficult to treat and representing one of the most significant barriers to functional recovery. One pathophysiologic pathway that may contribute to these alterations in reward circuitry in schizophrenia is inflammation. Increased inflammation has been reliably linked to deficits in reward processing and decreased motivation via effects of inflammatory cytokines on regions of the basal ganglia, including the ventral striatum. Previous findings show that some patients with schizophrenia reliably exhibit elevated concentrations of inflammatory markers and that inflammatory cytokines may be related to negative symptoms including decreased motivation. Relevant to the impact of inflammation on insulin signaling, measures of insulin sensitivity are significantly worse in patients with schizophrenia, including at illness onset. Moreover, antipsychotic medications lead to metabolic syndrome, contributing to risk for insulin resistance and ultimately diabetes. Insulin resistance is believed to be caused by increased inflammation, and in turn can contribute to inflammation through alterations in glucose metabolism.

This study uses an oral glucose tolerance test to test the hypothesis that insulin resistance drives inflammation. The researchers will recruit subjects with a range of insulin resistance, as measured by the Homeostatic Model Assessment of Insulin Resistance (HOMA-IR). This will allow the researchers to investigate the contributions of metabolic dysfunction and inflammation on inflammatory and metabolic markers, brain reward circuitry, motivational deficits, and negative symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to give written informed consent
* A primary diagnosis of schizophrenia, per the Diagnostic and Statistical Manual of Mental Disorders-5 (DSM-5), or schizoaffective disorder as diagnosed by the Mini International Neuropsychiatric Interview (MINI) 7.0
* Mini Mental Status Examination Score ≥24
* Brief Negative Symptom Scale Score ≥25
* No psychotropic medication changes for one month prior to study enrollment; may be taking other psychotropic non-antipsychotic medications (i.e., antidepressants, mood stabilizers, benzodiazepines)

Exclusion Criteria:

* Evidence of untreated or poorly controlled endocrine, thyroid, cardiovascular, hematological, renal, neurological disease, hepatitis B or C or HIV
* Current HbA1C ≥ 8.5%
* Prior treatment with antiviral or immunomodulatory drugs, including corticosteroids within six months of study entry
* Current treatment with antibiotics
* Primary diagnosis of major depressive disorder or bipolar disorder
* Active abuse of alcohol or illicit/prescription drugs within the past 6 months including a urine toxicology screen positive for drugs of abuse (patients may still be included with a positive tetrahydrocannabinol (THC) result at the discretion of the PI)
* Predominant left-handedness excluded for portions of the MRI scan
* Wide Range Achievement Test-3 Reading Scale (WRAT-3) score indicating less than 8th grade reading level, unless otherwise approved by the PI or PI's designee
* Any other condition which in the opinion of the investigator would make the patient unsuitable for enrollment, or could interfere with participating in or completing the protocol
* History of central nervous system trauma or active seizure disorder requiring medication
* Positive pregnancy test
* Presence of metal in the body (excludes from MRI scan only)
* Active suicidal ideation as determined by the PI and/or study staff
* Diagnosis of diabetes mellitus

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2020-08-31 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2022-03-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Goldsmith, MD, Principal Investigator — Emory University
Locations (6):
- United States (6):
  - Emory University Department of Psychiatry and Behavioral Sciences, Atlanta, Georgia
  - Grady Health System (non-CRN), Grady Health System (CRN), Ponce Center, Atlanta, Georgia
  - Emory Clinic, Emory University Hospital, Atlanta, Georgia
  - Emory University Clinical Research Network, Atlanta, Georgia
  - Emory University, Atlanta, Georgia
  - Emory Universtiy, Atlanta, Georgia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from Grady Health System in Atlanta, Georgia, USA. Participant enrollment began August 31, 2020, and all follow-up was complete by March 1, 2022.
Pre-assignment Details: This was an optional substudy underpowered to identify relationships between changes in inflammatory and metabolic markers pre- and post-OGTT with reward circuitry or motivational deficits. These analyses are thus exploratory and would serve as preliminary data for future research proposals.
Period: Overall Study
Arm/Group | Oral Glucose Tolerance Test (OGTT)
Started | 12
Completed | 11
Not Completed | 1
Not completed — Exclusion due to positive UDS (THC) test | 1

BASELINE CHARACTERISTICS:
Population: Participants who met all screening requirements.
Arm/Group | Oral Glucose Tolerance Test (OGTT)
Number analyzed (Participants) | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 11
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.36 (12.42)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 7
  White | 4
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 11

OUTCOME MEASURES:

1. Primary Outcome: Effort-Expenditure for Rewards Task (EEfRT) Score
Description: EEfRT is a multitrial game task assessing motivation in which participants choose between 2 different task difficulty levels to obtain monetary rewards. For all trials, participants make repeated manual button presses which raises the level of a virtual ''bar'' viewed onscreen by the participant. Participants are eligible to win the money allotted for each trial if they raise the bar to the ''top''. Each trial presents subjects with a choice between 'high effort' and 'low effort' tasks that require different amounts of button pressing. Reward magnitudes for the high-effort task vary between amounts, while reward magnitudes for the low-effort task remain constant. Trials also vary in terms of 3 levels of probability of winning the amount associated with the choice selected. The first 50 trials are used for analysis. Percentage of hard-task choices across all levels of probability is calculated from all hard choices. Lower percentages of hard task choices indicate decreased motivation.
Time Frame: Baseline, Hour 1
Measure: Mean (Standard Deviation); unit: proportion of hard-task choices
Arm/Group | Oral Glucose Tolerance Test (OGTT)
Number analyzed (Participants) | 11
proportion of hard-task choices
  Baseline | 0.268 (0.217)
  Hour 1 | 0.189 (0.153)

2. Secondary Outcome: Finger Tapping Task (FTT) Score
Description: The Finger Tapping Task (FTT) uses a specially adapted tapper that the subject is asked to tap as fast as possible. The subject is given 5 consecutive 10-second trials for the preferred and non-preferred hands.The FTT is design to assess subtle motor impairment and found to be altered in subjects with basal ganglia disorders and lesions. The finger tapping score is the mean number of taps of 5 trials and is computed for each hand.
Time Frame: Baseline, Hour 1
Population: 11 participants analyzed for baseline, but only 10 completed the 1-hour measurements. One participant could not complete the tasks for the left hand.
Measure: Mean (Standard Deviation); unit: number of taps on a 10 second counter
Arm/Group | Oral Glucose Tolerance Test (OGTT)
Number analyzed (Participants) | 11
number of taps on a 10 second counter
  Right Hand Baseline | 44.22 (6.74)
  Right Hand- Hour 1: number analyzed (Participants) | 10
  Right Hand- Hour 1 | 42.68 (11.44)
  Left hand Baseline | 39.98 (10.91)
  Left hand- Hour 1: number analyzed (Participants) | 10
  Left hand- Hour 1 | 42.01 (6.40)

3. Secondary Outcome: Trail Making Test Part A (TMT-A) Score
Description: The Trail Making Test-A is a timed task that provides information on motor function and speed of processing. In Part A of the TMT participants connect circles labeled with numbers, in ascending order. The score is the amount of time it takes for the participant to complete the task. The average time it takes to complete the task is 29 seconds and times longer than 78 seconds suggest a deficiency.
Time Frame: Baseline, Hour 1
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | Oral Glucose Tolerance Test (OGTT)
Number analyzed (Participants) | 11
Seconds
  Baseline | 38.86 (15.44)
  Hour 1 | 37.02 (16.12)

4. Secondary Outcome: Digit Symbol Substitution Task (DSST) Score
Description: The DSST is a subtest of the Wechsler Adult Intelligence Scale and involves graphimotor speed, visual scanning and memory, with about half of the variance being accounted for by graphimotor speed, a third by visual scanning and 4-5% by memory. Performance on the Digit Symbol Test has been found to correlate with subcortical (caudate) atrophy in disorders involving the basal ganglia. Respondents match symbols to numbers using a key presented at the top of the test page. The score is the number of correctly entered symbols in the given time period and higher scores indicate better performance.
Time Frame: Baseline, Hour 1
Measure: Mean (Standard Deviation); unit: Number of correct entered symbols
Arm/Group | Oral Glucose Tolerance Test (OGTT)
Number analyzed (Participants) | 11
Number of correct entered symbols
  Baseline | 60.55 (20.28)
  Hour 1 | 55.09 (20.98)

5. Secondary Outcome: Profile of Mood States (POMS) Brief Score
Description: The POMS is a 30-item rating scale designed to measure mood states across short periods. The POMS assess six mood factors: Tension-Anxiety, Depression-Dejection, Anger-Hostility, Vigor-Activity, Fatigue-Inertia, and Confusion-Bewilderment. Each item is rated on a 5-point scale where 0 = not at all and 4 = extremely. Total scores range from 0 to 120 and lower scores indicate a better state of mood.
Time Frame: Baseline, Hour 1
Population: Only participants with available data are included in the analysis. Baseline data was inadvertently lost and only available for two (2) participants.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Oral Glucose Tolerance Test (OGTT)
Number analyzed (Participants) | 11
Score on a scale
  Baseline: number analyzed (Participants) | 2
  Baseline | 37.50 (37.48)
  1 hour post | 20.27 (12.36)

6. Other Pre Specified Outcome: Fasting Blood Glucose
Description: Fasting blood glucose will be assessed to determine the impact of insulin resistance on inflammatory markers.
Time Frame: Baseline, Hours 1, 2, and 3
Population: Only baseline values were analyzed. Blood samples for exploratory outcome measures were not analyzed due to lack of funding.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Oral Glucose Tolerance Test (OGTT)
Number analyzed (Participants) | 11
mg/dL | 94.27 (18.78)

7. Other Pre Specified Outcome: Fasting Blood Insulin
Description: Fasting blood insulin will be assessed to determine the impact of insulin resistance on inflammatory markers.
Time Frame: Baseline, Hours 1, 2, and 3
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: mIU/L
Arm/Group | Oral Glucose Tolerance Test (OGTT)
Number analyzed (Participants) | 11
mIU/L | 12.9 (10.05)

8. Other Pre Specified Outcome: Neural Response to Reward Motivation Assessed by fMRI-adapted Version of the EEfRT
Description: Assessment of effort-based decision-making will be made using the EEfRT task adapted for fMRI. During each trial, subjects are presented with a choice between two levels of task difficulty, a High Effort option, and a Low Effort option. Unlike in the behavioral version of the task, subjects will not be required to make button presses during the scan. The reward magnitude for a No Effort option remains constant, while the reward magnitude for the High Effort option varies. Additionally, the amount of effort required for the High Effort option will vary between 20%, 50%, 80%, and 100% of the subject's maximum effort (set for each individual before the scan).
Time Frame: Baseline, Hour 3
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Change in Neural Response to Anticipating and Receiving Monetary Rewards Assessed by Monetary Incentive Delay (MID) Task
Description: Assessment of reward anticipation will be achieved using the MID task, conducted during functional MRI (fMRI) neuroimaging. Briefly, during this task participants have the opportunity to win or lose money by making a rapid button press in response to a target visual stimulus. The primary epoch of interest is the "anticipatory delay" - a period of ~2000ms that occurs after participants have been informed how much money they can win or lose on a given trial, but prior to the presentation of the target. This epoch has repeatedly been associated with robust ventral striatal activity. Participants will complete 2 functional runs of between 50 and 200 trials each (the number of trials will be decided at the discretion of the PI), with evenly distributed reward magnitudes.
Time Frame: Baseline, Hour 3
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Change in Cambridge Neuropsychological Test Automated Battery (CANTAB) Reaction Time Score
Description: This reaction time test includes simple and choice reaction time tasks and is divided into 5 stages requiring increasingly complex chains of responses and providing a distinction between reaction (or decision) time and movement latencies. Movement times on the CANTAB reaction time task have been slowed during interferon-alpha (IFN-α) treatment and correlated with IFN-alpha-induced depression and fatigue.
Time Frame: Baseline, Hour 1
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Plasma C-reactive Protein (CRP) Levels
Description: Plasma CRP will be assessed to determine the impact of insulin resistance on inflammatory markers.
Time Frame: Baseline, Hours 1, 2, and 3
Population: One participant did not get CRP drawn. Only the baseline sample was analyzed. Blood samples for exploratory outcome measures were not analyzed due to lack of funding.
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Oral Glucose Tolerance Test (OGTT)
Number analyzed (Participants) | 10
mg/L | 3.83 (4.67)

12. Other Pre Specified Outcome: Change in Monocyte Chemoattractant Protein-1 (MCP-1) Levels
Description: Fluorokine MAP Multiplex Human Biomarker Panels will be used to measure plasma inflammatory markers that have been found to be altered in schizophrenia. MCP-1 levels before and after the OGTT will be examined.
Time Frame: Baseline, Hours 1, 2, and 3
Population: Blood samples for exploratory outcome measures were not analyzed due to lack of funding.
Arm/Group | Oral Glucose Tolerance Test (OGTT)
Number analyzed (Participants) | 0

13. Other Pre Specified Outcome: Change in Interleukin-10 (IL-10) Levels
Description: Fluorokine MAP Multiplex Human Biomarker Panels will be used to measure plasma inflammatory markers that have been found to be altered in schizophrenia. IL-10 levels before and after the OGTT will be examined.
Time Frame: Baseline, Hours 1, 2, and 3
Population: Blood samples for exploratory outcome measures were not analyzed due to lack of funding.
Arm/Group | Oral Glucose Tolerance Test (OGTT)
Number analyzed (Participants) | 0

14. Other Pre Specified Outcome: Change in Soluble Interleukin-6 Receptor (sIL-6R) Levels
Description: Fluorokine MAP Multiplex Human Biomarker Panels will be used to measure plasma inflammatory markers that have been found to be altered in schizophrenia. sIL-6R levels before and after the OGTT will be examined.
Time Frame: Baseline, Hours 1, 2, and 3
Population: Only the baseline sample was analyzed. Blood samples for exploratory outcome measures were not analyzed due to lack of funding.
Arm/Group | Oral Glucose Tolerance Test (OGTT)
Number analyzed (Participants) | 0

15. Other Pre Specified Outcome: Change in Interleukin-6 (IL-6) Levels
Description: Fluorokine MAP Multiplex Human Biomarker Panels will be used to measure plasma inflammatory markers that have been found to be altered in schizophrenia. IL-6 levels before and after the OGTT will be examined.
Time Frame: Baseline, Hours 1, 2, and 3
Population: Blood samples for exploratory outcome measures were not analyzed due to lack of funding.
Arm/Group | Oral Glucose Tolerance Test (OGTT)
Number analyzed (Participants) | 0

16. Other Pre Specified Outcome: Change in Soluble TNF Receptor 2 (sTNFR2) Levels
Description: Fluorokine MAP Multiplex Human Biomarker Panels will be used to measure plasma inflammatory markers that have been found to be altered in schizophrenia. sTNFR2 levels before and after the OGTT will be examined.
Time Frame: Baseline, Hours 1, 2, and 3
Population: Blood samples for exploratory outcome measures were not analyzed due to lack of funding.
Arm/Group | Oral Glucose Tolerance Test (OGTT)
Number analyzed (Participants) | 0

17. Other Pre Specified Outcome: Change in Interleukin-1beta (IL-1beta) Levels
Description: Fluorokine MAP Multiplex Human Biomarker Panels will be used to measure plasma inflammatory markers that have been found to be altered in schizophrenia. IL-1beta levels before and after the OGTT will be examined.
Time Frame: Baseline, Hours 1, 2, and 3
Population: as for outcome 14
Arm/Group | Oral Glucose Tolerance Test (OGTT)
Number analyzed (Participants) | 0

18. Other Pre Specified Outcome: Change in Interleukin-1 Receptor Antagonist (IL-1RA) Levels
Description: Fluorokine MAP Multiplex Human Biomarker Panels will be used to measure plasma inflammatory markers that have been found to be altered in schizophrenia. IL-1RA levels before and after the OGTT will be examined.
Time Frame: Baseline, Hours 1, 2, and 3
Population: Blood samples for exploratory outcome measures were not analyzed due to lack of funding.
Arm/Group | Oral Glucose Tolerance Test (OGTT)
Number analyzed (Participants) | 0

19. Other Pre Specified Outcome: Change in Tumor Necrosis Factor (TNF)-Alpha Levels
Description: Fluorokine MultiAnalyte Profiling (MAP) Multiplex Human Biomarker Panels will be used to measure plasma inflammatory markers that have been found to be altered in schizophrenia. TNF-alpha levels before and after the OGTT will be examined.
Time Frame: Baseline, Hours 1, 2, and 3
Population: Blood samples for exploratory outcome measures were not analyzed due to lack of funding.
Arm/Group | Oral Glucose Tolerance Test (OGTT)
Number analyzed (Participants) | 0

20. Other Pre Specified Outcome: Change in Resting State Scan
Description: For the resting state and task-based functional connectivity analysis, whole brain, subject-level correlation maps indicating regional similarity with the striatal seed region time series will be generated and Fisher transformed to Z-score maps. In addition, data reduction strategies will be employed to address inflammatory marker collinearity in analyses combining relevant inflammatory markers. To assess the significance of correlated activity with each bilateral seed region, paired t-tests will be conducted on participants' Z-score maps, adjusted for multiple comparisons. For significant brain regions, descriptive statistics will be used to characterize the mean, standard deviation, and standard error of the Z scores.
Time Frame: Baseline, Hour 3
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Information on adverse events was collected beginning at the time of consent to participate in the study throughout study participation up to 10 days.
Arm/Group | Oral Glucose Tolerance Test (OGTT)
All-Cause Mortality (participants affected / at risk) | 0/11
Serious Adverse Events (participants affected / at risk) | 0/11
Other Adverse Events (participants affected / at risk) | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-01-31): https://cdn.clinicaltrials.gov/large-docs/16/NCT03818516/Prot_SAP_001.pdf
  • Informed Consent Form (2023-02-15): https://cdn.clinicaltrials.gov/large-docs/16/NCT03818516/ICF_002.pdf